CLINICAL TRIAL: NCT02098616
Title: RHACE 1: Rapid HepAtitis C Elimination Trial - A Pilot Evaluation of Twice Daily Fixed Dose Combination Asunaprevir +Daclatasvir + BMS-791325 ± Weight Based Ribavirin in Treatment-Naïve, Non-cirrhotic Patients With Chronic Genotype 1a Hepatitis-C for Eight, Six or Four Weeks
Brief Title: Rapid Hepatitis C Elimination Trial- A Pilot Study of Daclatasvir/Asunaprevir/BMS-791325 With or Without Ribavirin To Treat Hepatitis C Virus
Acronym: RHACE 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Morgan, MD (Other)
Collaborators: VA Long Beach Healthcare System (U.S. Federal Agency); National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Timothy Morgan, MD, Chief, Hepatology, Southern California Institute for Research and Education
Organization: Southern California Institute for Research and Education (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #1285; AI443-128 (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; RNA Virus Infections; Antiviral Agents; Drug Resistance, Viral
MeSH Terms: conditions — Hepatitis C; Hepatitis; Hepatitis, Chronic; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; RNA Virus Infections | interventions — daclatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day for 8 weeks
  Interventions: Drug: DCV/ASV/BMS-791325
- Arm 2 (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day for 6, 8 or 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325
- Arm 3 (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day for 4 weeks
  Interventions: Drug: DCV/ASV/BMS-791325
- Arm A (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day plus weight based ribavirin orally twice a day for 8 weeks
  Interventions: Drug: DCV/ASV/BMS-791325 + RBV
- Arm B (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day plus weight based ribavirin orally twice a day for 6, 8 or 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325 + RBV
- Arm C (Experimental): Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day plus weight based ribavirin orally twice a day for 4 weeks
  Interventions: Drug: DCV/ASV/BMS-791325 + RBV

INTERVENTIONS:
Drug: DCV/ASV/BMS-791325 — Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) orally twice a day
  Other Names: Fixed Dose Combination (FDC) of Daclatasvir/Asunaprevir/BMS-791325
  Arms: Arm 1; Arm 2; Arm 3
Drug: DCV/ASV/BMS-791325 + RBV — Fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg and BMS-791325 75 mg) tablet orally twice a day plus weight based ribavirin orally twice a day
  Arms: Arm A; Arm B; Arm C

SUMMARY:
The purpose of this study is to determine whether treatment with Daclatasvir/Asunaprevir/BMS-791325, with or without ribavirin, for 8, 6, or 4 weeks is feasible for the treatment of genotype 1a chronic hepatitis C in patients without cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1a
* HCV RNA ≥ 10,000 IU/mL at screening
* Treatment-naïve subjects with no previous exposure to an interferon formulation (ie, IFNα, pegIFNα), ribavirin (RBV), or HCV direct acting antiviral (DAA; protease, polymerase inhibitor, etc.)

Exclusion Criteria:

* Evidence of cirrhosis
* Liver or any other organ transplant
* Current or known history of cancer within 5 years prior to enrollment
* Documented or suspected hepatocellular carcinoma (HCC)
* Not eligible for sofosbuvir + pegylated interferon + ribavirin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response | Post treatment week 12
  Proportion of treated subjects in each enrolled arm with sustained virologic response (SVR)12. SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) target detected or target not detected (TD/TND) at post treatment Week 12

SECONDARY OUTCOMES:
Safety | Up to end of treatment (+7 days)
  On treatment safety, as measured by frequency of serious adverse events (SAEs) and adverse events (AEs), discontinuations due to AEs, and rates and grades of select laboratory abnormalities including liver function tests and hematology laboratory abnormalities in each arm
Sustained virologic response | 2, 4 and 24 weeks post-treatment
  Proportion of treated subjects in each arm with SVR2, SVR4 and SVR 24, defined as HCV RNA < lower limit of quantification (LLOQ) target detected or target not detected (TD/TND) at post treatment Weeks, 2, 4, and 24 respectively
Post treatment virologic response | post treatment Weeks 2 (SVR2), 4 (SVR4), and 24 (SVR24)
  To assess the proportion of subjects who achieve sustained virologic response (SVR) 2, SVR4 and SVR24.
On treatment virologic response | On-treatment Day 2 and Weeks 1, 2, 4, 6, 8 and 12
  To assess antiviral activity, as measured by the proportion of subjects who achieve HCV RNA <lower limit of detection (LLOD) and/or < lower limit of quantification (LLOQ) at each on treatment visit.
Virologic failure | On-treatment Day 2 and Weeks 1, 2, 4, 6, 8 and 12 and Post Treatment Weeks 2, 4, 12 and 24
  To assess the proportion of subjects with virologic failure (including on treatment virologic breakthrough and relapse) and evaluate the emergence of viral resistant mutations.
Day 2 positive predictive value | Post treatment Week 12
  To assess the predictive value of Day 2 virologic response on sustained virologic response (SVR) 12
Interferon lambda genotype and virologic response | On-treatment Day 2 and Weeks 1, 2, 4, 6, 8 and 12 and Post Treatment Weeks 2, 4, 12 and 24
  To compare the virologic response of subjects by genotype for interferon (IFN) lambda variants [' IL28B' and IFNL4-ΔG]

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R. Morgan, MD, Principal Investigator — VA Long Beach Healthcare System/Southern California Institute for Research and Education
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States